CLINICAL TRIAL: NCT05538637
Title: Reliability and Accuracy of Mitral Velocity Time-integral Variability With Passive Leg Raising as a Marker of Preload-responsiveness in Patients With Acute Circulatory Failure in the ICU.
Brief Title: Is Mitral Velocity Time-integral a Marker of Preload-responsiveness in Patients With Acute Circulatory Failure?
Status: Completed | Type: Observational
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Professor of Anesthesiology and Intensive Care Medicine - Head of surgical intensive care unit, Avicenna Military Hospital
Other Study IDs: Mitral VTI ICU-AMH
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Preload-responsiveness
Keywords: preload-responsiveness; acute circulatory failure; left ventricular outflow tract velocity time integral; mitral valve velocity time integral; echocardiography
MeSH Terms: conditions — Shock | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Mitral velocity time-integral variability measurement before and after passive leg raising.
  Mitral velocity time-integral variability measurement after fluid loading in preload-responsiveness patients.
  Other Names: Mitral velocity time-integral variability

SUMMARY:
The aim of this is to assess the reliability of the variability of the mitral velocity time-integral with passive leg raising to predict the fluid responsiveness in patients with acute circulatory failure in intensive care.

DETAILED DESCRIPTION:
Adult patients with acute circulatory failure will be included in the study. An initial echocardiography is performed in patients placed in a semi-recumbent position. On the apical views (4 and 5-chamber views), the left ventricular outflow tract velocity time integral (LVOT-VTI) and mitral valve (MV-VTI) velocity time integral are measured (baseline values). Then a passive leg raise test is performed and the parameters (LVOT-VTI and MV-VTI) are measured again. Preload-responsiveness is defined by an increase in LVOT-VTI of at least 10%. In preload-responsive patients, a fluid loading with 500 ml of 0.9% saline administered over 15 minutes is performed. Immediately after fluid therapy, the same parameters are recorded during a third echocardiography. An increase of 10% or more of LVOT-VTI , compared with baseline, defines fluid responsiveness. Patients are monitored using the standard of care practices. Hemodynamic assessment includes repetitive echocardiographic examinations if needed. In patients with shock, invasive blood pressure is monitored with an arterial catheter.

ELIGIBILITY:
Inclusion Criteria: Acute circulatory failure.

Exclusion Criteria:

* Recent surgery (<5 days)
* Suspected or confirmed intra-abdominal hypertension.
* Intracranial hypertension.
* Severe mitral valve disease: Severe mitral insufficiency or severe mitral stenosis
* Acute cor pulmonale
* Atrial fibrillation
* Low echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute circulatory failure, with or without arterial hypotension. Acute circulatory failure is defined by the presence of signs of tissue hypoperfusion : prolonged capillary refil time (>5 seconds), mottling, acrocyanosis, oliguria (<0.5 mL/kg/h for more than an hour), altered mental status, lactate>2 mmol/l or metabolic acidosis (pH<7.35, base excess >-5). Arterial hypotension is defined by systolic blood pressure (SBP) < 90mmHg, mean arterial pressure (MAP) < 65 mmHg or a drop in SBP ≥ 40 mmHg. Shock is defined by the association of an acute circulatory failure and arterial hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Reliability and accuracy of the change in mitral valve velocity time-integral (cm) to discriminate preload-responsiveness | through study completion, an average of 6 months
  Reliability and accuracy of the change in mitral valve velocity time-integral (cm) measured by echocardiography (before and after passive leg raising) to discriminate preload-responsive patients.
Reliability and accuracy of the change in mitral valve velocity time-integral (cm) to discriminate fluid-responsiveness | through study completion, an average of 6 months
  Reliability and accuracy of the change in mitral valve velocity time-integral (cm) measured by echocardiography (before and after fluid loading with 500 ml of saline) to discriminate fluid-responsive patients.

CONTACTS AND LOCATIONS:
Overall Officials: Younes Aissaoui, MD, Principal Investigator — Cadi Ayyad University. Faculty of Medicine and Pharmacy. Avicenna Military Hospital.
Locations (1):
- Avicenna Military Hospital, Marrakesh, Marrakesh Tensift El Haouz, Morocco

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion for 2 years
Access Criteria: healthcare workers

REFERENCES:
- [Derived] Aissaoui Y, Jozwiak M, Bouchama A, Bennjakhoukh H, Bencharfa B, Didi M, Abouqal R, Belhadj A. Evaluation of the mitral velocity-time integral changes induced by a passive leg raising test as a marker of fluid responsiveness in critically ill patients. J Clin Monit Comput. 2025 Dec;39(6):1159-1168. doi: 10.1007/s10877-025-01320-z. Epub 2025 Jul 8. PMID 40627255